CLINICAL TRIAL: NCT04416633
Title: A Prospective, Multicenter, Phase-IV Clinical Trial to Assess Safety of Durvalumab in Indian Adult Patients With Locally Advanced, Unresectable Non-small Cell Lung Cancer (NSCLC)
Brief Title: Study to Access Safety of Durvalumab in Indian Adult Patients With Locally Advanced NSCLC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D133HC00003
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Unresectable Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab (Other): Single arm, Durvalumab , IV
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — 500-mg/120-mg IV

SUMMARY:
A prospective, multicenter, Phase-IV clinical trial to assess safety of Durvalumab in Indian adult patients with locally advanced, unresectable non-small cell lung cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent prior to any study specific Procedures
2. Male or female aged 18 years or older
3. As per local prescribing information and in view of positive benefit-risk assessment, patient prescribed Durvalumab treatment as per independent clinical judgment of treating physician for either

Exclusion Criteria:

1. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study
2. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drug, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
3. Prior exposure to any anti-PD-1 or anti-PD-L1 antibody including durvalumab.
4. For NSCLC cohort only:

   1. Mixed small cell and non-small cell lung cancer histology
   2. Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy.
   3. Patients with ≥Grade 2 pneumonitis from prior chemoradiation therapy
5. Active or prior documented autoimmune disease within the past 2 years, inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis), primary immunodeficiency, organ transplant that requires therapeutic immunosuppression, hypersensitivity to study drug or any excipient, leptomeningeal carcinomatosis, tuberculosis.

   NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
6. Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
7. Any condition that, in the opinion of the investigator, would interfere with evaluation of the study drug or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Faridabad
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, Mohali
  - Research Site, Mumbai
  - Research Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D133HC00003_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HC00003&attachmentIdentifier=83ec647c-7105-458b-b475-50c9aca1dded&fileName=D133HC00003_CSP_Redacted.pdf&versionIdentifier=
- See also: D133HC00003_SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HC00003&attachmentIdentifier=ee66849b-39d9-4728-b7cf-900ae62b6aad&fileName=D133HC00003_SAP_Redacted.pdf&versionIdentifier=
- See also: D133HC00003_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HC00003&attachmentIdentifier=70767b06-31e7-4396-83cf-7948ecd0e888&fileName=D133HC00003_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Durvalumab: Durvalumab administered intravenously for over 60 minutes at 10 mg/kg every 2 weeks.
  The treatment period for this study was 20 weeks, which corresponded to 10 doses of study drug administration.
Period: Overall Study
Arm/Group | Durvalumab
Started | 100
Completed | 69
Not Completed | 31
Not completed — Death | 1
Not completed — Disease progression as per investigator's clinical and imaging assessment | 17
Not completed — AE greater than Grade 3 related to study drug | 1
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set
Arm/Group | Durvalumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.04 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 82
Race/Ethnicity, Customized [Number; unit: Participants]
  INDIAN | 100
  OTHER | 0
Height [Mean (Standard Deviation); unit: centimeters] | 164.44 (9.04)
Weight [Mean (Standard Deviation); unit: kilograms] | 61.12 (11.69)

OUTCOME MEASURES:

1. Primary Outcome: Number and Proportion of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI)
Description: The number and proportion of participants who experienced AEs, SAEs, and AESIs, including interstitial lung disease/pneumonitis-like events and on-study deaths are presented.
Time Frame: Evaluation Phase (Day 1 to 141) to Follow-up Phase (90 days after End of Evaluation Visit [Day 141])
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: All the patients who are enrolled in the study and received at least one dose of an investigational product as an IV infusion
Arm/Group | Safety Population
Number analyzed (Participants) | 100
Participants
  Any Adverse Event | 74
  Any Serious Adverse Event | 21
  Any Treatment Emergent Adverse Event | 74
  Any Serious Treatment Emergent Adverse Event | 21
  Treatment Emergent Adverse Event related to IMP | 26
  Treatment Emergent Adverse Event leading to IMP discontinuation | 13
  Treatment Emergent Adverse Event leading to Death | 4
  Adverse events of special interest | 8

2. Primary Outcome: Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI)
Description: The number of events of AEs, SAEs, and AESIs, including interstitial lung disease/pneumonitis-like events and on-study deaths are presented.
Time Frame: Evaluation Phase (Day 1 to 141) to Follow-up Phase (90 days after End of Evaluation Visit [Day 141])
Measure: Number; unit: events
Arm/Group | Safety Population
Number analyzed (Participants) | 100
events
  Any Adverse Event | 267
  Any Serious Adverse Event | 27
  Any Treatment Emergent Adverse Event | 250
  Any Serious Treatment Emergent Adverse Event | 27
  Treatment Emergent Adverse Event related to IMP | 55
  Treatment Emergent Adverse Event leading to IMP discontinuation | 24
  Treatment Emergent Adverse Event leading to Death | 4
  Adverse events of special interest | 8

ADVERSE EVENTS:
Time Frame: Day 1 to Day 230 of the Follow-up Period (ie, up to 8 months).
Description: Adverse events were to be reported by the participant(or, when appropriate, by a caregiver, surrogate, or the patient's legally authorized representative).
  The investigator and any designees were responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE.
Arm/Group | Durvalumab
All-Cause Mortality (participants affected / at risk) | 4/100
Serious Adverse Events (participants affected / at risk) | 21/100
Other Adverse Events (participants affected / at risk) | 69/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=100)
Death (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Autoimmune myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=100)
Constipation (Gastrointestinal disorders) | 4 (5)
Pallor (Vascular disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 5 (5)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Fatigue (General disorders) | 4 (4)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 19 (20)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Amylase increased (Investigations) | 6 (6)
Blood thyroid stimulating hormone abnormal (Investigations) | 1 (3)
Blood uric acid increased (Investigations) | 1 (1)
Crystal urine present (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 4 (5)
Weight increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (26)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 12 (13)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT04416633/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04416633/SAP_001.pdf